CLINICAL TRIAL: NCT06411652
Title: The Effect of Foot Reflexology and Therapeutic Touch on Fatigue, Depression and Quality of Sexual Life in Women Receiving Hemodialysis Treatment
Brief Title: The Effect of Foot Reflexology and Therapeutic Touch on Fatigue, Depression and Quality of Sexual Life in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, CANSU AĞRALI, Research Assistant at the Midwifery Department of the Faculty of Health Sciences, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OsmaniyeKAU-SBF-CA-02
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: Women Health
MeSH Terms: conditions — Depression | interventions — Musculoskeletal Manipulations; Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Experimental model with pretest posttest control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reflexology Group (Experimental): The researcher has received a practitioner reflexology certificate. The researcher will begin the massage during the second hour of dialysis, as the patient's condition is more stable and the unit is less crowded due to routine care. Before the intervention, the patient's privacy will be protected in the reflexology group; The researcher will sit in a chair at the foot of the patient's bed and perform a reflexology massage.
  Interventions: Other: Reflexology
- Therapeutic Touch Group (Experimental): In order to perform Therapeutic Touch application, the researcher attended the first level training prepared by the International Therapeutic Touch Association and received a certificate. For therapeutic touch application, the researcher will start the application in the second hour of dialysis, as the patient's condition is more stable and the unit is less crowded due to routine care. Therapeutic touch application will be applied to women in the hemodialysis care unit, twice a week for four weeks, for a total of 8 sessions, each lasting 15 minutes.
  Interventions: Other: Therapeutic Touch
- Control group (No Intervention): No intervention will be made.

INTERVENTIONS:
Other: Reflexology — 1. First, the patient's foot will be cleaned with cotton dipped in warm water,
  2. In order not to disturb the patient, the hands will be warmed and one or two ccs of baby oil will be used to facilitate the massage.
  3. Before applying the main technique, the first two minutes of each session will be spent using the relaxation technique, which involves back and forth movements with the palm of the palm on the outer edge of the foot, from the outer part of the ankle to the little toe, to relieve muscle tension and spasm.
  4. Then, alternate pressure will be applied to the reflex points of the right thumb by taking the heel of one foot in the left hand.
  Arms: Reflexology Group
Other: Therapeutic Touch — 1. The procedure will be explained to the woman,
  2. The procedure will be performed in the patient's bed.
  3. The practitioner will center by making his body, mind and emotions quiet and focused, prepare himself for the practice and remain centered throughout the intervention,
  4. There will be good intentions to help the woman get treatment,
  5. In order to scan the energy field, the patient's entire body will be held with the palms of the practitioner's hands facing the patient, it will be moved with a soft movement from
  Arms: Therapeutic Touch Group

SUMMARY:
This study aims to examine the effects of foot reflexology and therapeutic touch on fatigue, depression and sexual quality of life in women receiving hemodialysis treatment. Hemodialysis treatment may have negative effects on the quality of sexual life and mental health of female patients. In this context, understanding the potential healing effects of foot reflexology and therapeutic touch on sexual health and fatigue and depression in these individuals may contribute to the development of more effective support and treatment strategies.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) stands out as a rapidly increasing important health problem globally. CKD is a universal public health priority associated with significantly higher morbidity and mortality and excessive health care costs. The most common form of renal replacement therapy is hemodialysis. In patients with chronic kidney disease treated with hemodialysis, the disappearance of the survival advantage of women over men in the general population deeply affects the life experience of women. Among the additional difficulties that women face in this process compared to men, the inability to maintain their emotional resilience, failure to comply with treatment, and failure to meet their social support needs come to the fore.

The problems caused by hemodialysis and chronic illness create a significant burden on women, both materially and spiritually, and negatively affect women's quality of life. Common and common conditions include sleep disorders, fatigue, depression and pain. In addition, higher levels of sexual dysfunction have been reported in women with hemodialysis, and it has been stated that loss of sexuality may reduce self-confidence and cause problems in marriage. Chronic hemodialysis patients, especially female patients, should be supported in terms of sexual dysfunctions and psychosocial conditions. Therefore, health professionals should evaluate the psychosocial lives of especially female patients and provide the necessary support. Health professionals' use of complementary approaches to reduce patients' problems and improve their negative emotional states increases the effectiveness of medical treatment.

Reflexology and therapeutic touch are among the low-cost and complication-free nursing interventions. These nursing interventions can be used together with medical treatments to reduce stress and balance the body. Studies indicate that reflexology application and therapeutic touch can be effective in improving sexual function and positive emotions. However, when the literature is examined, it is observed that there are no studies evaluating therapeutic touch intervention in women receiving hemodialysis treatment, and reflexology studies are quite inadequate. Therefore, our study aims to examine the effects of foot reflexology and therapeutic touch on fatigue, depression and sexual quality of life in women receiving hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being sexually active
* Volunteering to participate in the research

Exclusion Criteria:

* The patient is 65 years or older or under 18 years of age
* Having a communication problem

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Sexual Quality of Life Scale-Female | Four Weeks
  Sexual Quality of Life Scale, Symonds et al. It is a scale whose validity and reliability have been established by. The scale is a scale that can be applied to all women over the age of 18, but the validity and reliability study of the original scale was conducted on women in the 18-65 age group. The scale is easy to apply, six-point Likert type, and consists of 18 items that individuals can answer on their own. Each item is expected to be answered considering your sexual life in the last four weeks. In the original version of the scale, it is stated that each item can be scored between 1-6 or 0-5. In this study, a 1-6 point system (1 = Completely agree, 2 = Largely agree, 3 = Partially agree, 4 = Partially disagree, 5 = Largely disagree, 6 = Strongly disagree) was used. In this way, the score range that can be obtained from the scale is between 18-108. It is accepted that as the score obtained from the scale increases, the individual's quality of sexual life also increases.

SECONDARY OUTCOMES:
Fatigue Severity Scale | Four Weeks
  The Fatigue Severity Scale, developed by Krup, is a scale consisting of nine items that evaluates the general impact of fatigue on daily activities. The Turkish validity and reliability of the scale was determined by Armutlu et al. Made by. In the scale, individuals are asked to rate the fatigue they felt throughout the past week on a scale from 1 to 7. Each section is scored between 1 (completely disagree) and 7 (completely agree). The total score is calculated by taking the average of nine items. The cut-off value for pathological fatigue was determined as 4 and above. The lower the total score, the less fatigue. Armutlu et al. In the study, it was stated that the Cronbach's alpha coefficient of the scale was 0.94.
Beck Depression Scale | Four Weeks
  This scale, which was first developed by Aaron T. Beck (1961), was adapted into Turkish in 1988 and its validity and reliability were checked by Hisli. Beck 21 depression scale consists of 21 items and each of these items has four options. Each item receives a score between 0 and 3, and a depression score is obtained by summing these scores. The highest total score that can be obtained is 63, and a high score indicates the severity of depression. The cut-off score was taken as 17. Those who scored 17 or more were considered to have symptoms of depression. In the validity and reliability study of BDI, the Cronbach α reliability coefficient was determined as 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Ağralı, Study Director — Osmaniye Korkut Ata University
Locations (1):
- Osmaniye New State Hospital, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No